CLINICAL TRIAL: NCT00741598
Title: The Efficacy and Safety of Galantamine for Dysfunction in Bipolar Disorder
Brief Title: Efficacy and Safety of Galantamine for Improving Dysfunction in People With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dan V. Iosifescu, M.D., M.Sc., Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 10-1060; R01MH079157 (NIH); 1R01MH079157-01A2 (NIH); DATR A5-ETMA
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine-ER (Experimental): Participants will receive treatment with extended release galantamine
  Interventions: Drug: Galantamine-ER
- Galantamine placebo (Placebo Comparator): Participants will receive treatment with placebo.
  Interventions: Drug: Galantamine placebo

INTERVENTIONS:
Drug: Galantamine-ER — Galantamine-ER 8 to 24 mg per day for 16 weeks
  Other Names: Razadyne-ER
  Arms: Galantamine-ER
Drug: Galantamine placebo — Galantamine placebo 8 to 24 mg per day for 16 weeks
  Other Names: placebo
  Arms: Galantamine placebo

SUMMARY:
This study will examine whether extended release galantamine, a drug approved by the Food and Drug Administration to reduce cognitive impairments in people with Alzheimer's disease, can perform the same function in stable people with bipolar disorder.

DETAILED DESCRIPTION:
Approximately 2.6% of Americans age 18 and older, or 5.7 million people, suffer from bipolar disorder. The manic and depressive episodes associated with bipolar disorder prevent normal functioning in individuals with the disorder, but functional impairment can occur even when bipolar disorder is in remission. Previous research indicates that this impairment in stable individuals with bipolar disorder is linked to neurocognitive deficits, such as problems with memory and attention. The drug extended release galantamine increases the level of acetylcholine, a neurotransmitter important for memory, available in the brain. This drug has already been approved by the FDA to treat neurocognitive impairment in Alzheimer's disease patients. This study will examine whether administering the drug to individuals with bipolar disorder who are in remission can also reduce their neurocognitive deficits and improve the quality of their life. The study will also examine the safety of the drug for use in the obsessive-compulsive disorder population.

Participation in this study will last about 18 weeks and will involve six study visits. Each of the first two visits will include 2 hours of clinical, physical, and self-report tests, the first for screening and the second to establish physical and mental health baseline measurements. Participants will then be randomly assigned to receive either galantamine or placebo daily for 16 weeks, and they will be provided with enough of the assigned pill to last until the next visit. Half hour visits on Weeks 4, 8, and 12 will consist of psychological self-report tests and interviews, clinical assessment of side effects from the drug, and the determination by the examining doctor and participant whether to increase, decrease, or maintain the same level of the drug. Participants will also be given enough of the drug to last until the next visit. The final visit, on Week 16, will last 2 hours and will consist of the same tests administered at the baseline visit in addition to the neuropsychological tests administered at the screening visit. The full range of tests will measure physical health, verbal memory, mental flexibility, attention, life impairment, and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Bipolar I disorder or Bipolar II disorder
* A baseline Hamilton-D 17 score of less than 10 at screening visit
* A baseline Young Mania Rating Scale (YMRS) score of less than 10 at screening visit
* No acute episodes of depression or mania for the previous 12 weeks
* Score of 17 or higher on the Massachusetts General Hospital (MGH) Cognitive and Physical Functioning Questionnaire
* Treated with psychiatric medications, alone or in combination, having only minimal, mild or moderate cognitive burden [as determined by a score of less than 3.5 on the MGH Cognitive Impact of Psychotropic Medications Scale (CIPMS).
* Able to understand English

Exclusion Criteria:

* DSM-IV diagnosis of Bipolar NOS, Cyclothymia, or Schizoaffective Bipolar type.
* Meets DSM-IV criteria for acute manic, depressive, or mixed bipolar episode or had met full criteria for 2 consecutive weeks within the past 12 weeks prior to assessment
* Treated with psychiatric medications with large effects on cognition (as determined by a MGH Cognitive Impact of Psychotropic Medications Scale score of 4.0 or above)
* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy)
* Serious suicide or homicide risk
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* History of seizure disorder, brain injury, or any known neurological disease (multiple sclerosis, degenerative disease such as ALS, Parkinson disease and any movement disorders, etc)
* The following DSM-IV diagnoses: 1) organic mental disorders; 2) any diagnosis of dementia; 3) substance use disorders, including alcohol, active within the last year; 4) schizophrenia; 5) delusional disorder; 6) psychotic disorders not elsewhere classified; 7) schizoaffective disorder; 8) major depressive disorder; 9) acute bereavement; 10) severe borderline or antisocial personality disorder
* Presence of mood congruent or mood incongruent psychotic features
* Clinical or laboratory evidence of hypothyroidism
* History of multiple adverse drug reactions, allergy to galantamine or other AChEIs
* Current use, or use within the last week, of excluded drugs (psychotropic medications and other central nervous system (CNS)-active drugs)
* Taken an investigational psychotropic drug within the last year
* Had electroconvulsive therapy (ECT) within the 6 months preceding enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan V. Iosifescu, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai & Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- See also: Click here for more information on the Massachusetts General Hospital's Bipolar Clinic and Research Program. — http://www.massgeneral.org/psychiatry/services/treatmentprograms.aspx?id=1132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study procedures were conducted between January 2009 and June 2015 at two sites: the Mood and Anxiety Disorders Program at Icahn School of Medicine at Mount Sinai and the Bipolar Clinical Research Program at the Massachusetts General Hospital.
Groups:
- Galantamine-ER: 16-week treatment with flexible doses (8-24mg/day)
- Placebo: placebo equivalent
Period: Overall Study
Arm/Group | Galantamine-ER | Placebo
Started | 33 | 39
Completed | 24 | 30
Not Completed | 9 | 9
Not completed — Lost to Follow-up | 3 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine-ER | Placebo | Total
Number analyzed (Participants) | 33 | 39 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (13.1) | 47.8 (12.3) | 46.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Scores on the California Verbal Learning Test (CVLT-II) at Screening and Week 16
Description: CVLT is a test measuring verbal learning and verbal memory. Subjects are expected to remember a list of words. They are asked to repeat the words remembered 5 times (5 trials). Each of the words correctly remembered, in each trial, is marked as 1 point. The outcome measures presented are:
  CVLT Total Trials 1-5, Baseline = Number of total words remembered, sum of trials 1-5, at baseline CVLT Total Trials 1-5, Week 16 = Number of total words remembered, sum of trials 1-5, at week 16.
Time Frame: Measured at screening and Week 16
Measure: Mean (Standard Deviation); unit: number of total words remembered
Groups:
- Placebo: 16-week treatment with flexible doses of placebo equivalent
Arm/Group | Galantamine-ER | Placebo
Number analyzed (Participants) | 24 | 30
number of total words remembered
  CVLT Total Trials 1-5, Baseline | 50.15 (13.36) | 47.21 (10.77)
  CVLT Total Trials 1-5, Week 16 | 58.88 (14.69) | 52.90 (13.17)

2. Primary Outcome: Scores on the Wisconsin Card Sorting Test (WCST) at Screening and Week 16
Description: WCST (Wisconsin Card Sorting Test) is a neuropsychological test measuring the ability to display flexibility in the face of changing schedules of reinforcement. Subjects are presented with cards and requested to match them. Unbeknownst to the subject, the matching rules change while the test is delivered. The test measures subjects' ability to understand the new rules.
  The outcome measures presented are Total correct baseline = total correct card choices at baseline Total errors baseline = total erroneous card choices at baseline Total correct week 16 = total correct card choices at week 16 Total errors baseline = total erroneous card choices at week 16
Time Frame: Measured at screening and Week 16
Measure: Mean (Standard Deviation); unit: number of card choices made
Arm/Group | Galantamine-ER | Placebo
Number analyzed (Participants) | 24 | 30
number of card choices made
  Total Correct Baseline | 45.87 (23.16) | 44.11 (19.69)
  Total Errors Baseline | 29.70 (19.38) | 29.79 (22.54)
  Total Correct Week 16 | 51.94 (23.79) | 44.28 (23.72)
  Total Errors Week 16 | 27.75 (18.52) | 29.61 (18.52)

3. Primary Outcome: The Conners' Continuous Performance Test (CPT) at Baseline, Weeks 4, 8, 12, and 16
Description: Conner's CPT (Conner's Continuous Performance Task) is a neuropsychological test that measures a person's sustained and selective attention. Subjects are instructed to click the space bar when they are presented with any letter except the letter "X". The person must refrain from clicking if they see the letter "X" presented. Clicking to the letter "X" is a commission error, not clicking to other letters are omission errors.
  The outcome measures presented are Total number of errors = Total number of omission + commission errors This outcome measure is presented at each study visit (baseline, week 4, week 8, week 12, and week 16)
Time Frame: Measured at screening; baseline; and Weeks 4, 8, 12, and 16
Measure: Mean (Standard Deviation); unit: total number of errors
Arm/Group | Galantamine-ER | Placebo
Number analyzed (Participants) | 24 | 30
total number of errors
  CPT Total omission + commission errors, Baseline | 22.16 (19.78) | 19.40 (12.38)
  CPT Total omission + commission errors, Week 4 | 21.87 (21.10) | 19.24 (18.08)
  CPT Total omission + commission errors, Week 8 | 15.61 (17.67) | 16.39 (11.15)
  CPT Total omission + commission errors, Week 12 | 9.91 (10.11) | 16.41 (14.70)
  CPT Total omission + commission errors, Week 16 | 14.23 (20.34) | 15.18 (12.20)

4. Secondary Outcome: The Range of Impaired Functioning Tool (LIFE-RIFT)
Description: The LIFE-RIFT is a brief measure of functional impairment. The total scale score is a sum of four items with range of scale from 0 to 26 (from no impairment to severe impairment).
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine-ER | Placebo
Number analyzed (Participants) | 24 | 30
units on a scale
  LIFE-RIFT total score, Baseline | 10.39 (2.52) | 9.41 (2.89)
  LIFE-RIFT total score, Week 4 | 9.66 (2.79) | 9.03 (2.42)
  LIFE-RIFT total score, Week 8 | 9.07 (2.80) | 8.53 (2.36)
  LIFE-RIFT total score, Week 12 | 8.24 (2.35) | 8.03 (2.80)
  LIFE-RIFT total score, Week 16 | 8.88 (3.19) | 8.20 (2.91)

5. Secondary Outcome: Quality of Life Satisfaction Questionnaire (Q-LES-Q)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-report instrument designed to measure the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. There are 16 areas of functioning, each scored from 1 (very poor) to 5 (very good). The range of scores is 16-80, with lower scores representing lower functioning and satisfaction.
  The outcome measures presented are Q-LES-Q Total score = Sum of all scores from all 16 areas of functioning
Time Frame: Screening
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine-ER | Placebo
Number analyzed (Participants) | 24 | 30
units on a scale
  Q-LES-Q Total, Baseline | 62.3 (9.79) | 63.03 (13.18)
  Q-LES-Q Total, Week 4 | 66.03 (15.00) | 64.75 (15.32)
  Q-LES-Q Total, Week 8 | 62.62 (12.34) | 65.28 (15.29)
  Q-LES-Q Total, Week 12 | 66.96 (10.32) | 66.52 (14.89)
  Q-LES-Q Total, Week 16 | 64.75 (9.98) | 61.31 (19.36)

ADVERSE EVENTS:
Arm/Group | Galantamine-ER | Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/39
Other Adverse Events (participants affected / at risk) | 32/33 | 39/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine-ER (N=33) | Placebo (N=39)
Trouble sleeping (General disorders) | 6 | 7
Drowsy (General disorders) | 5 | 8
Nervous/Hyper (General disorders) | 2 | 2
Fatigue (General disorders) | 3 | 6
Irritable (General disorders) | 3 | 4
Headache (General disorders) | 6 | 5
Nausea/vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes